CLINICAL TRIAL: NCT04122014
Title: Effectiveness of an Exercise Program to Improve Balance and Dual Task in Hemophilic Patients. Clinical Trial
Brief Title: Exercise Program to Improve Balance in Hemophilic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Felipe Querol Fuentes, Principal Investigator, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H20190326180948
Record Dates: First submitted 2019-07-24; First posted 2019-10-10 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Usual daily activities
  Interventions: Other: Normal daily activities
- Training group (Experimental): Each subject will participate in 2 sessions each week during 3 months.
  Interventions: Other: Progressive balance training

INTERVENTIONS:
Other: Progressive balance training — Progressive balance training program
  Arms: Training group
Other: Normal daily activities — Usual daily activities
  Arms: Control group

SUMMARY:
This study evaluates the effectiveness of a program of physiotherapy exercises to train the balance and dual task in adults patients with hemophilia

DETAILED DESCRIPTION:
The objective of the study is to create an exercise program to improve the static and dynamic balance in hemophilic patient. In addition, the effect of the exercise program on dual task, functionality, proprioception, QoL, risk of falls and the kinesiophobia will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of haemophilia A or B
* Willingness to exercise twice a week during the training program and to complete the pre- and post-program evaluations
* Approval by their hematologist to participate in the exercise program
* With hemostatic coverage supervised by your hematologist.
* Age between 18 and 60 years
* Informed consent signed.

Exclusion Criteria:

* Non adherence to instruction on proper exercise technique
* Surgical procedures performed 6 months prior to or during the exercise program
* A major bleeding episode that posed a risk or prevented exercise
* Need for major surgery
* Suffer from dizziness
* Withdrawal of informed consent
* Acquired hemophilia

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change of postural balance: amplitude of Center of Pressure (CoP) displacements | baseline and 3 months
  Amplitude of CoP displacements will be assessed in millimeters using a computerized balance system. Higher displacements indicate worse balance.
Change of postural balance: velocity of Center of Pressure (CoP) displacements | baseline and 3 months
  Velocity of CoP displacements will be assessed in millimeters using a computerized balance system. Higher velocity indicate worse balance.
Change of postural balance: sway area of Center of Pressure (CoP) displacements | baseline and 3 months
  Sway area of CoP displacements will be assessed in mm^2 using a computerized balance system. Higher sway area indicate worse balance.
Change of dual task balance: amplitude of Center of Pressure (CoP) displacements | baseline and 3 months
  Amplitude of CoP displacements will be assessed in millimeters using a computerized balance system. Patient will perform a cognitive task (e.g. counting) while maintaining balance. Higher displacements indicate worse balance.
Change of dual task balance: velocity of Center of Pressure (CoP) displacements | baseline and 3 months
  Velocity of CoP displacements will be assessed in millimeters using a computerized balance system. Patient will perform a cognitive task (e.g. counting) while maintaining balance. Higher velocity indicate worse balance.
Change of dual task balance: sway area of Center of Pressure (CoP) displacements | baseline and 3 months
  Sway area of CoP displacements will be assessed in mm^2 using a computerized balance system. Patient will perform a cognitive task (e.g. counting) while maintaining balance. Higher sway area indicate worse balance.

SECONDARY OUTCOMES:
Limits of Stability (LOS): success rate | baseline and 3 months
  Evaluations will be done by NedSVE/IBV balance platform. Indices: Max Excursions (%), Directional Control (%), Success (%), LOS rate (%) will be recorded during forward, backward, right and left side movements.
Limits of Stability (LOS): time | baseline and 3 months
  Evaluations will be done by NedSVE/IBV balance platform. Indices: Reaction Time (s), Confinement Time (s), will be recorded during forward, backward, right and left side movements.
The Berg Balance Scale | baseline and 3 months
  Balance will be assessed with the Berg Balance Scale (BBS), a 14-item physical performance measure of static and dynamic balance found to be reliable. Scoring ranges from 0-56, with higher scores indicating better balance. A score of <46 identifies an individual at risk for falls after stroke.
Functional capacity: The Timed "Up & Go" test | baseline and 3 months
  Timed "Up & Go" will be used to measure functional capacity. It is a simple test used to assess a person's mobility and requires both static and dynamic balance. Less time to complete the test in seconds implies better outcome.
Functional capacity: Sit-to-stand test | baseline and 3 months
  Sit-to-stand test (3 repetitions) will be used to measure functional capacity. Less time to complete the test in seconds implies better outcome.
Functional capacity: 2-minutes walk test | baseline and 3 months
  Evaluation of functional capacity during walking by using 2 minutes walk test. More distance covered in 2 minutes implies better outcome.
Haemophilia Activities List (HAL) | baseline and 3 months
  The Haemophilia Activities List questionnaire measures the impact of hemophilia on self-perceived functional abilities in adults.
  It contains 42 multiple choice questions in seven domains:
  Lying/sitting/kneeling/standing (8 items) Functions of the legs (9 items) Functions of the arms (4 items) Use of transportation (3 items) Self-care (5 items) Household tasks (6 items) Leisure activities and sports (7 items) The most important outcomes are the overall sum score and three component scores relating to upper extremity activities, basic lower extremity activities, and complex lower extremity activities. The score is obtained using a Likert scale with 5 options: always=2, mostly=3, sometimes=4, rarely=5 and never=6 (complemented by the option "impossible=1" for those people who can not perform such activity). Subscales are summed, with a total score from 0- 252 and higher values represent a worse outcome (greater self-perceived difficulty in carrying out the activities).
Functional Independence Scale for Hemophilia (FISH) | baseline and 3 months
  Observed activity limitations will be measured with the Functional Independence Scale for Hemophilia (FISH) as part of the Activity Domain.
  The scale studies 8 activities (eating and grooming, bathing, dressing, chair, squatting, walking, stairs and running), which are classified into the three groups (Self care, Transfers and Locomotion) and their score ranges from 1 - 4 (1 being the highest dependency and 4 being the greatest independence to perform the exercises). Subscales are summed, with a total score from 8-32 and higher values represent a better outcome.
  The FISH has been validated for use in developing countries. It consists of observed activities of daily living that are scored for quality.
Quality of Life related with health: questionnaire | baseline and 3 months
  Measured by a Specific questionnaire for Quality of Life related with health evaluation for adults with haemophilia (A36Haemophilia-QoL), which explores 9 areas. Subscales and score range: Physical health: 0-32; Daily activities: 0-16; Joints: 0-12; Pain: 0-8; Treatment satisfaction: 0-8; Difficulties treatment: 0-16; Emotional functioning: 0-20; Mental health: 0-12; Social activity: 0-20. Subscales are summed, with a total score from 0-144 and higher values represent a better outcome (more Quality of Life perceived).
Kinesiophobia | baseline and 3 months
  Kinesiophobia will be evaluated by Tampa Scale for Kinesiophobia (TSK-11SV) (Spanish adaptation. Gómez-Pérez, López-Martínez y Ruiz P., 2011). Scoring: Items are summed, with a total score from 11-44 and higher values represent a worse outcome (more pain interference in behavior).
Modified Falls Efficacy Scale (mFES) | baseline and 3 months
  MFES is a 14-item questionnaire related to daily indoor and outdoor physical activities. It is a 10-point visual analog scale of confidence level in completing a particular activity (item) without falling, rated from 0 to 10, where 0 denotes not confident or sure at all, and 10 denotes completely confident or sure. The total score for the 14 items ranges from 0 to 140.
Joint health status | baseline
  Joint clinical evaluation of elbows, knees and ankles by using The Hemophilia Joint Health Score 2.1 (HJHS). The full score range goes from 0 to 124 points (0-20 points for each of the six joints evaluated, plus 4 points for the overall assessment of gait. 0 means no joint damage, whereas the higher the value, the higher the degree of arthropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Querol-Fuentes, MD, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chimeno-Hernandez A, Perez-Alenda S, Cruz-Montecinos C, Carrasco JJ, Aguilar-Rodriguez M. Multimodal Exercise Program of Balance and Strength Improves Dynamic Balance, Strength and Functionality and Decreases the Risk of Falls in Adults With Haemophilia. Haemophilia. 2025 May;31(3):544-556. doi: 10.1111/hae.70040. Epub 2025 Mar 28. PMID 40153408